CLINICAL TRIAL: NCT01606280
Title: Reporting of Amyloidosis Stem Cell Transplantation Outcomes
Brief Title: Long-term Outcomes of Patients With Primary Amyloidosis After Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Morie Gertz, principal investigator, Mayo Clinic
Other Study IDs: 11-005003
Record Dates: First submitted 2012-03-15; First posted 2012-05-25 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Amyloidosis
Keywords: Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examines the value of stem cell transplantation in managing light chain amyloidisis.

DETAILED DESCRIPTION:
1. How does age at diagnosis affect prognosis in primary amyloidosis?
2. How do lab values at diagnosis such as Creatinine, AST/ALT, total serum protein, serum gamma globulin/immunoglobulin levels affect prognosis in primary amyloidosis?
3. How does degree of organ involvement/number of organs involved affect prognosis in primary amyloidosis?
4. How does initial treatment affect prognosis in primary amyloidosis?

4. How do the specifics the stem cell transplant protocol affect prognosis in primary amyloidosis?

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Stem cell transplantation less than age 75

Exclusion Criteria:

* Creatinine > 3.0
* BNP > 10000

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient receiving transplantation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Survival | up to 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States